CLINICAL TRIAL: NCT06579352
Title: Intermediate Size Expanded Access Study of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSC) In Patients With Duchenne Muscular Dystrophy
Brief Title: Expanded Access Study of UC-MSC in DMD Patients
Status: Available | Type: Expanded Access
Sponsor: MED Institute Inc. (Industry)
Collaborators: Signature Biologics (Unknown)
Responsible Party: Sponsor
Other Study IDs: IND 16561 - Serial 0017
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Human Umbilical Cord Mesenchymal Stem Cells (UC-MSC) — Umbilical cord-derived mesenchymal stem cells administered intravenously.

SUMMARY:
The primary objective of this study is to provide UC-MSC treatment to patients with DMD.

Secondary objectives will be to further evaluate treatment-related adverse events as well as changes in DMD-related functional testing/assessments, blood laboratories, and inflammation related biomarker levels over time.

DETAILED DESCRIPTION:
The study will enroll ambulatory male participants between the ages of 5 and 10, who will receive four, 3-day intravenous dose cycles of UC-MSC treatment, each administered every three months. Participants will be closely monitored throughout the study period for treatment-related adverse events and changes in DMD-related functional assessments at specific follow-up intervals through 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male sex by birth with a genetically confirmed diagnosis of Duchenne Muscular Dystrophy (DMD).
2. Age is greater than or equal to 5 and less than or equal to 10 years.
3. Has a North Star Ambulatory Assessment (NSAA) score greater than 13 and less than 30.
4. Demonstrates the ability to perform the "time to rise" test in under 10 seconds.
5. Is up-to-date on immunizations.
6. Is on a stable dose of glucocorticoids for at least 12 weeks prior to study participation, except for weight-based or toxicity-related adjustments.
7. Is on a stable dose of supplements for at least 12 weeks prior to study participation.
8. Has the ability to comply with the requirements of the study and the ability to understand and provide written informed assent and a guardian's consent.
9. Patient must be either a non-responder to or a poor candidate for treatment with another established therapy.

Exclusion Criteria:

1. Active cancer or prior diagnosis of cancer within the past year (patients with basal and squamous cell cancer of the skin will not be excluded).
2. BMI > 45 kg/m².
3. Any other condition (including concomitant treatment) that, in the judgment of the Investigator or Sponsor, would be a contraindication to enrollment, study product administration (e.g., known hypersensitivity to dimethyl sulfoxide (DMSO), Human Serum Albumin (HSA), or PlasmaLyte), or follow-up.
4. Treatment with an exon skipping therapy within 3 months of study start.
5. Cognitive delay or impairment that can confound motor development in the opinion of the investigator.
6. Major surgery within 3 months prior to Day 0 or planned surgery or procedures that could affect the conduct of the study.

Ages: 5 Years to 10 Years | Sex: Male
Age Groups: Child
Gender Based: Yes — Study participants will be ambulatory males aged 5-10 with genetically confirmed DMD.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Rare Disease Center, Denton, Texas, United States